CLINICAL TRIAL: NCT03388086
Title: Comparing the Efficacy of Two Doses of Onabotulinum Toxin for the Treatment of Neurogenic Detrusor Overactivity - a Retrospective Cohort Study
Brief Title: Efficacy of Two Onabotulinum Toxin Doses
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2017-17
Record Dates: First submitted 2017-12-13; First posted 2018-01-02 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Neurogenic Bladder; Overactive Detrusor
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Onabotulinum 300 units
  Interventions: Drug: Injection of Onabotulinum toxin
- Onabotulinum 200 units
  Interventions: Drug: Injection of Onabotulinum toxin

INTERVENTIONS:
Drug: Injection of Onabotulinum toxin — multiple injections of Onabotulinum toxin into the detrusor muscle

SUMMARY:
The changes in bladder function after the injection of Onabotulinum toxin into the detrusor in individuals with neurogenic bladder overactivity will be investigated retrospectively. The records of all patients treated with Onabotulinum toxin injections into the detrusor since 2000 will be evaluated. The changes in the urodynamic values after the injection of 300 units of Onabotulinum toxin will be compared with the changes after the injection of 200 units. Furthermore, the differences in urinary continence, duration between injections, side effects and complications between the two groups will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic detrusor overactivity
* spinal cord injury
* Onabotulinum toxin injections into the detrusor from 2000-2017

Exclusion Criteria:

* missing urodynamic values before or after Onabotulinum toxin injections

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with Onabotulinum toxin for neurogenic detrusor overactivity as a result of spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
change in detrusor pressure post-injection | within 3 months before injection; within 2 months after injection
  bladder detrusor pressure during storage phase

SECONDARY OUTCOMES:
maximum bladder volume | within 3 months before injection; within 2 months after injection
bladder compliance | within 3 months before injection; within 2 months after injection
  The relationship between a change in bladder volume and the change in detrusor pressure (ΔDV/ΔDP).
reflexive bladder volume | within 3 months before injection; within 2 months after injection
complications | within 2 months after injection
presence of urinary incontinence | within 3 months before injection; within 2 months after injection

OTHER OUTCOMES:
lesion level | at the time of spinal cord injury
lesion severity | at the time of spinal cord injury
method of bladder evacuation | within 2 months after injection
  evacuation by intermittent catheterization, reflex voiding, suprapubic catheter , electric stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland